CLINICAL TRIAL: NCT02458261
Title: Pharmacokinetics and Pharmacodynamics of Extended-Infusion Cefepime in Continuous Renal Replacement Therapy
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Carri Philpott, Pharmacist, UC Health, UCMC, University of Cincinnati
Other Study IDs: 2014-6119
Record Dates: First submitted 2015-04-27; First posted 2015-06-01 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Drug Mechanism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples that are being collected are as follows: serum, continuous renal replacement therapy effluent, and urine (if patient is making urine during sample collection). Drug assays will be performed for each sample and samples will be disposed of after the final analysis is complete. The assays are not interventional and patient care does not change as a result of study enrollment.
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective, multi-center study aims to determine the pharmacokinetics and pharmacodynamics of extended-infusion cefepime in continuous renal replacement therapy (CRRT).

DETAILED DESCRIPTION:
This prospective, multi-center study aims to determine the pharmacokinetics and pharmacodynamics of extended-infusion cefepime in CRRT. Patients on CRRT who are being initiated on cefepime 2000 mg IV every eight hours with a four-hour infusion will be considered for enrollment. Pre- and post-membrane serum levels will be drawn at scheduled intervals for both the first dose and again during another dose at steady state. Concomitant effluent and urine levels will also be obtained. A pharmacokinetic analysis will be performed and Monte Carlo simulations will be used to determine the probability of target attainment for various pharmacodynamic endpoints. Documented organism MICs will be used to determine the cumulative fraction of response.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to medical intensive care unit (MICU), surgical intensive care unit (SICU), neuroscience intensive care unit (NSICU), or cardiovascular intensive care unit (CVICU), at the University of Cincinnati Medical Center, or the mixed ICU at West Chester Hospital
* Patients receiving continuous venovenous hemofiltration or continuous venovenous hemodialysis
* Receiving empiric or definitive cefepime 2 g IV every 8 hours with a four-hour infusion

Exclusion Criteria:

* Prisoners
* Pregnant women
* Patients with cystic fibrosis
* Burns patients
* 24-hour urine output > 400 mL or unknown

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients on continuous renal replacement therapy who are being initiated on cefepime 2000 mg IV every 8 hours with a four-hour infusion
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Composite pharmacokinetic and pharmacodynamic profile of extended-infusion cefepime in CRRT | up to 12 months
  Each patient will have samples collected on both the first dose and another dose at presumed steady state (dose four, five, or six) to determine the pharmacokinetic and pharmacodynamic profile of extended-infusion cefepime in CRRT. Pharmacokinetic outcomes calculated include half life, volume of distribution, and area under the plasma concentration versus time curve. Sieving and saturation coefficients will also be calculated as appropriate. Time above the minimum inhibitory concentration will be the primary pharmacodynamic outcome studied.

IPD SHARING:
Plan to Share IPD: Undecided